CLINICAL TRIAL: NCT07046481
Title: Functional Capacity, Physical Activity, Health-related Quality of Life and Fatigue in Young Cancer Survivors, 5-10 Years After Diagnosis
Brief Title: Physical Activity and Quality of Life in Childhood Cancersurvivors- a Long-term Follow-up
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Registration was withdrawn from clinicaltrials.gov as the ISRCTN registry was found to be more suitable for our study.
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1162 SUS S&D; 2023-06785-01 (Other: EPM)
Record Dates: First submitted 2024-12-08; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Leukemia, Acute; Brain Neoplasms; Physical Fitness; Quality of Life; Fatigue
Keywords: physical activity; physical function; rehabilitation; inactivity; pediatric
MeSH Terms: conditions — Leukemia; Brain Neoplasms; Fatigue; Motor Activity; Sedentary Behavior | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This is a feasiblity study of the intervention Physical Activity on Prescription. Participants who are inactive according to the WHO recommendations, will be recruited to the study. Pre and post intervention assessment will be compared and participant's notes in a personal activity diary will be analyzed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical activity on prescription (Experimental): World Health Organization recommends that children should engage in moderate to vigorous physical activity for at least 60 minutes a day. Participants who in the cross-sectional study are found not to fulfill the WHO recommendation on physical activity, will be recruited to the study where physical activity will be prescribed and performed according to the preferences of the participant.
  Pre and post intervention physical activity, physical function, health related quality of life and fatigue will be assessed using standardized measures.
  Interventions: Other: Physical activity

INTERVENTIONS:
Other: Physical activity — One or two physical activities according to the participant´s preferences will be selected and prescribed and specified for frequence and intensity. The selected activity/-ies could be of any type, as long as they increase the heart rate. The activity/-ies should be performed regularly during 12 weeks, A training diary will be used to monitor and register the activities.

SUMMARY:
The project intends to study physical functional capacity and degree of physical activity health related quality of life and fatigue. Also, we aim to study if the Physical Activity on Prescription (PAP) intervention is a useful method among physically inactive childhood cancer survivors to increase level of activity.

The questions the study aim to answer:

* What is the physical functional capacity, degree of physical activity, health related quality of life and fatigue among childhood cancer survivors 5- 10 yars after dignosis?
* Is the Physical Activity on Prescription intervention feasible for physically inactive childhood cancer survivors and what effect do they experience in terms of physical functioning, physical activity, sedentary behavior, fatigue and health-related quality of life?

Participants aged 5-17 years who have been treated for leukemia or brain tumor will be invited to participate. Physical functional capacity and degree of physical activity are assessed with standardized assessment instruments by a physiotherapist. Prior to the visit, participants are also asked to complete questionnaires on HRQoL and fatigue.

Participants identified as physically inactive are offered to participate in a PAP intervention. Functional ability scores from previous studies are used as a baseline and are supplemented with objective measurements of physical activity and followed up after the intervention.

DETAILED DESCRIPTION:
The challenges of childhood cancer survivors to incorporate exercise and physical activity into their lives need to be systematically studied so that health care professionals can provide adequate support during and after treatment. It is therefore of great clinical relevance to gather knowledge on how physiotherapists can design and support regular physical activity and exercise for childhood cancer survivors. The project intends to study the feasibility of the PAP intervention on physical functioning, physical activity, sedentary behavior, fatigue and health-related quality of life among physically inactive children and adolescents who have survived childhood cancer, and whether it is a suitable method for these patient groups.

Methodology Participants must have been treated for brain tumor or acute lymphoblastic leukemia and be eligible for follow-up at the Pediatric Department at Skåne University Hospital before the age of 18.

Physical functioning, level of physical activity/sedentary behavior, health-related quality of life and fatigue are studied in a descriptive cross-sectional study. All children and adolescents aged 5-17 years treated for leukemia or brain tumor and scheduled for their usual follow-up 5-10 years after diagnosis identified using registers from (Swedish national registry of long-term follow-up in childhood cancer) SALUB are invited to participate, the sample is consecutive over a three-year period. Assessments of physical functioning and physical activity are performed by a physiotherapist in conjunction with a visit to the pediatric clinic. Prior to the visit, participants will complete the questionnaires on health related quality of life and fatigue.

Participants identified as physically inactive according to the WHO guidelines will be recruited to the intervention study where the PAP will be offered.

The intervention study explores the feasibility of benefits and effects on physical functioning, physical activity/ sedentary behavior, fatigue and health related quality of life after a PAP intervention in physically inactive childhood cancer survivors in a feasibility study. Participants identified as physically inactive in the initial study are invited to participate.

Data collection from the cross sectional study will be used as baseline and supplemented with objective measurements of physical activity using an accelerometer before the start of the three-month intervention. Participants will be allowed to choose one or two physical activities. The activity can either be an organized sport activity or an everyday task such as walking the dog or cycling to school. To facilitate the selection of an activity that the participants are motivated to perform, a standardized survey is conducted. During the intervention, participants complete an exercise diary regarding intensity and frequency but also other experiences related to the activity. Motivational interviewing is used to support participants to make changes in their physical activity level. At the end of the intervention, levels of physical activity, sedentary behavior, physical functioning, health-related quality of life and fatigue and accelerometer measurements are compared to baseline measurements.

The total number of participants treated for brain tumor or leukemia and available for screening of inactivity over a three-year period corresponds to about 50-55 and 70 persons respectively. This means that in total there will be approximately 120 participants to invite to the screening study. Participants will be included until the total number of participants reaches 50. Those who are inactive will be recruited to the intervention study, where physical activity on prescription will be used in order to increase the participant's activity level. We estimate that twenty participants may be eligible for participating.

The study is descriptive in nature, so a power calculation cannot be performed.

Importance of the project The project will increase knowledge about young cancer survivors' functional capacity, physical activity level, health-related quality of life and prevalence of fatigue. In addition, the need for rehabilitative interventions will be identified, knowledge will be deepened on how physical activity can be promoted for young cancer survivors and how this can affect the individual's future functional capacity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with Acute Lymphatic Leukemia or brain tumor 5- 10 years ago and available for follow-up at Lund University hospital.

Exclusion Criteria:

* Unable to walk with assistive devices, unable to communicate in the Swedish language

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Bruiniks Oseretsky test of motor proficiency | Assessments will be performed prior to the 12 week-intervention and directly after finishing the intervention.
  BOT-2 measures fine and gross motor proficiency, with subtests that focus on stability, mobility, strength, coordination, and object manipulation. The test is tailored to school-aged children and young adults among the ages of 4-21 years, who have varying motor control abilities ranging from normal to mild or moderate. The BOT-2 provides several types of derived scores that assists in interpreting performance. Scale scores (mean = 15, standard deviation = 5), confidence intervals, age equivalents, and descriptive categories are used to describe subtest performance. Standard scores (mean = 50, standard deviation = 10), confidence intervals, percentile ranks, and descriptive categories are used to describe composite and Short Form performance.

SECONDARY OUTCOMES:
6 minut- walk test | Assessments will be performed prior to the 12 week-intervention and directly after finishing the intervention.
  The test is a submaximal excercise test used to assess aerobic capacity and endurance. The distance covered over a 6 minutes is used as the outcome by which to compare changes in performance capacity. The patient is instructed to continoiusly walk in a self-selected speed between two cones 30 m apart during 6 minutes. The patient is monitored for heart rate and oxygen saturation during the test and will be asked to assess level of excersion using the Borg Breathlessness scale.
  The longer distance walked the better result.
Grippit | Assessments will be performed prior to the 12 week-intervention and directly after finishing the intervention.
  Isometric grip strength is measured with the Grippit instrument, a electronic device used clinically that registers the grip force (N) generated by the muscles. Grippit consists of an elliptical handle, 12.5 cm in circumference, an electronic unit and an adapter for connection to electricity. The grip handle and a forearm support are fixed on a board, which enables the test position to be standardised. Higher force imply better grip strength.
Canadian Occupational Performance Measure | Assessments will be performed prior to the 12 week-intervention and directly after finishing the intervention.
  The Canadian Occupational Performance Measure is an outcome measure designed to capture a client's self-perception of performance in everyday living, over time. The COPM measures performance and satisfaction in self-care, productivity and leisure from the client's perspective and is rated from 1- 10 where a higher score imply that the client is more satisfied with performance with the specifified activity.
Pediatric Quality of Life | Assessments will be performed prior to the 12 week-intervention and directly after finishing the intervention.
  The PedsQL Measurement Model is a modular approach to measuring health-related quality of life (HRQOL) in healthy children and adolescents and those with acute and chronic health conditions. Following dimensions are assessed:
  Physical Functioning , Emotional Functioning , Social Functioning , School Functioning. Results are presented in Summary Scores; Total Scale Score, Physical Health Summary Score and Psychosocial Health Summary Score. Items are reversed scored and linearly transformed to a 0-100 scale, so that higher scores indicate better HRQOL
Pediatric Quality of Life Multifatigue scale | Assessments will be performed prior to the 12 week-intervention and directly after finishing the intervention.
  The PedsQL™ Multidimensional Fatigue Scale is a specific module of the PedsQL™ and was designed as a generic symptom-specific instrument to measure fatigue in patients with acute and chronic health conditions as well as healthy school and community populations. The module includes 18 items to be scored between 0-4, result may vary between 0-71 where a higher scores imply less fatigue.
International physical activity questionnaire | Assessments will be performed prior to the 12 week-intervention and directly after finishing the intervention.
  The International Physical Activity Questionnaire (IPAQ) can be used to obtain comparable estimates of physical activity. It was designed for physical activity surveillance and can be used with care in other contexts. Standardized assessment to survey the patients self assessed level of activity and inactivity during the last 7 days.
  The IPAQ result in the amount of minutes of diffrerent levels of activity, the more minutes the patient is active in higher levels of activity the better.
Accelerometer | Assessments will be performed prior to the 12 week-intervention and directly after finishing the intervention.
  The patient will wear a device to measure and record movement during seven consequtive days. Information on the amount, frequency and duration of physical activity will be collected and analyzed using a computer soft-ware by the researchers. Result will be presented in minutes at different levels of activity, the higher amount of minutes in higher levels of activity the more active.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Brogårdh, Prof, Study Director — Department of health Sciences, Medical faculty, Lund University. Sweden

IPD SHARING:
Plan to Share IPD: Yes
All de-identified IPD that underlie results in the publication
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Result] Hagstromer M, Oja P, Sjostrom M. The International Physical Activity Questionnaire (IPAQ): a study of concurrent and construct validity. Public Health Nutr. 2006 Sep;9(6):755-62. doi: 10.1079/phn2005898. PMID 16925881
- [Result] Varni JW, Burwinkle TM, Katz ER, Meeske K, Dickinson P. The PedsQL in pediatric cancer: reliability and validity of the Pediatric Quality of Life Inventory Generic Core Scales, Multidimensional Fatigue Scale, and Cancer Module. Cancer. 2002 Apr 1;94(7):2090-106. doi: 10.1002/cncr.10428. PMID 11932914
- [Result] Lauruschkus K, Hallstrom I, Westbom L, Tornberg A, Nordmark E. Participation in physical activities for children with cerebral palsy: feasibility and effectiveness of physical activity on prescription. Arch Physiother. 2017 Nov 28;7:13. doi: 10.1186/s40945-017-0041-9. eCollection 2017. PMID 29340207
- [Result] Dinas PC, Koutedakis Y, Flouris AD. Effects of exercise and physical activity on depression. Ir J Med Sci. 2011 Jun;180(2):319-25. doi: 10.1007/s11845-010-0633-9. Epub 2010 Nov 14. PMID 21076975
- [Result] Slater ME, Steinberger J, Ross JA, Kelly AS, Chow EJ, Koves IH, Hoffmeister P, Sinaiko AR, Petryk A, Moran A, Lee J, Chow LS, Baker KS. Physical Activity, Fitness, and Cardiometabolic Risk Factors in Adult Survivors of Childhood Cancer with a History of Hematopoietic Cell Transplantation. Biol Blood Marrow Transplant. 2015 Jul;21(7):1278-83. doi: 10.1016/j.bbmt.2015.04.007. Epub 2015 Apr 10. PMID 25865649
- [Result] Han JW, Kim HS, Hahn SM, Jin SL, Shin YJ, Kim SH, Lee YS, Lee J, Lyu CJ. Poor bone health at the end of puberty in childhood cancer survivors. Pediatr Blood Cancer. 2015 Oct;62(10):1838-43. doi: 10.1002/pbc.25581. Epub 2015 May 13. PMID 25970742
- [Result] Landier W, Armenian S, Bhatia S. Late effects of childhood cancer and its treatment. Pediatr Clin North Am. 2015 Feb;62(1):275-300. doi: 10.1016/j.pcl.2014.09.017. Epub 2014 Oct 18. PMID 25435123
- [Result] Moody K, Meyer M, Mancuso CA, Charlson M, Robbins L. Exploring concerns of children with cancer. Support Care Cancer. 2006 Sep;14(9):960-6. doi: 10.1007/s00520-006-0024-y. Epub 2006 Apr 26. PMID 16639553
- [Result] Cox CL, Montgomery M, Oeffinger KC, Leisenring W, Zeltzer L, Whitton JA, Mertens AC, Hudson MM, Robison LL. Promoting physical activity in childhood cancer survivors: results from the Childhood Cancer Survivor Study. Cancer. 2009 Feb 1;115(3):642-54. doi: 10.1002/cncr.24043. PMID 19117349
- [Result] Ness KK, Leisenring WM, Huang S, Hudson MM, Gurney JG, Whelan K, Hobbie WL, Armstrong GT, Robison LL, Oeffinger KC. Predictors of inactive lifestyle among adult survivors of childhood cancer: a report from the Childhood Cancer Survivor Study. Cancer. 2009 May 1;115(9):1984-94. doi: 10.1002/cncr.24209. PMID 19224548
- See also: World Health Organization's guidelines on physical activity and sedentary behaviour. — https://apps.who.int/iris/bitstream/handle/10665/337001/9789240014886-eng.pdf